CLINICAL TRIAL: NCT04685538
Title: A Prospective, Observer-masked, Randomized Clinical Trial to Investigate and Compare the Clinical Efficacy of Chloroprocaine 3% Gel and Tetracaine 0.5% Eye Drop as Topical Anestheticsin Phacoemulsification.
Brief Title: Chloroprocaine 3% Gel Eye Drop as Topical Anestheticsin Phacoemulsification.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sintetica SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHL.3/01-2019/M
Record Dates: First submitted 2020-12-15; First posted 2020-12-28 (Actual); Results first posted 2022-10-27 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2021-04

CONDITIONS: Cataract
Keywords: Cataract; Eye; Chloroprocaine
MeSH Terms: conditions — Cataract | interventions — DMAC2L protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chloroprocaine 3% (Experimental): All the eligible patients will be administrated by Chloroprocaine 3 % according to the randomization criteria.
  Interventions: Drug: Chloroprocaine 3%
- Tetracaine 0.5% (Active Comparator): All the eligible patients will be administrated by Tetracaine 0.5% according to the randomization criteria.
  Interventions: Drug: Tetracaine 0.5%

INTERVENTIONS:
Drug: Chloroprocaine 3% — Administration: three IMP drops instillation as follow:
  * 1st Drop instillation, then wait for 5 minutes
  * Eye Disinfection, then wait for 2 minutes
  * 2nd Drop instillation, then wait for 1 minute
  * 3rdDrop instillation, then wait for 1 minute
  * Start of Surgery.
  Other Names: Arm 1
  Arms: Chloroprocaine 3%
Drug: Tetracaine 0.5% — Administration: three IMP drops instillation as follow:
  * 1st Drop instillation, then wait for 5 minutes
  * Eye Disinfection, then wait for 2 minutes
  * 2nd Drop instillation, then wait for 1 minute
  * 3rdDrop instillation, then wait for 1 minute
  * Start of Surgery.
  Other Names: Arm 2
  Arms: Tetracaine 0.5%

SUMMARY:
Randomized clinical trial, multicenter, two-armed, to investigate and compare the clinical efficacy of chloroprocaine 3% gel and tetracaine 0.5% eye drop as topical anestheticsin phacoemulsification. This prospective, observer masked, randomised, controlled, equivalence phase 3 study will be conducted in approximately 4 European Countries. Sintetica intends to perform a phase 3 study on patients undergoing cataract surgery to assess the safety and efficacy of topical anaesthesia using chloroprocaine gel.

DETAILED DESCRIPTION:
Prospective,randomized, multi-center, active-controlled, masked-observer, parallel-group, competitive equivalence study. The study has been designed to assess the equivalence of chloroprocaine 3% gel (Test) with respect to tetracaine 0.5% solution (Reference) in surface anesthesia. Patients in both groups will receive three drops of study products before surgery. The study will include a Selection visit (Day -90/Day -1), an Inclusion visit (Day 1/surgery day), a Follow-up visit (Day 2, phone visit), a Final visit (Day 8), and a Follow-up phone call - Optional (Day 28, phone visit).

Selection visit (Visit 1, Day -90/Day -1):

Patients scheduled to undergo cataract surgery in a single eye will be informed about the aims, procedures and possible risks of the study and will be asked to sign the informed consent form for the inclusion in the trial.

Inclusion visit/Surgery (Visit 2, Day 1):

Before the anesthesia, patients will be questioned about previous and concomitant ocular and non-ocular treatments. Inclusion /exclusion criteria and patient status will be verified. Patients will be randomized to either chloroprocaine 3% gel (Test) or tetracaine 0.5% eye drop (Reference) treatment group.

Follow-up visit/phone visit (Visit 3, Day 2):

Concomitant ocular and non-ocular treatments, AEs, and patient global satisfaction will be assessed.

Final visit (Visit 4, Day 8 ± 1 day):

Concomitant ocular and non-ocular treatments, ocular symptoms, best far corrected visual acuity in both eyes, endothelial cell count, corneal thickness, blood pressure and heart rate, and AEs will be assessed. Slit lamp examination and fluorescein test, IOP in both eyes, and fundoscopy will be performed.

Optional visit/phone visit (Visit 5, Day 28 ± 3 days):

Concomitant ocular and non-ocular treatments and AEs resolution will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent
2. Male or female aged≥ 18 years
3. Senile or pre-senile cataract
4. Scheduled to undergo cataract surgery in a single eyeat a time (clear corneal self-sealing incisions - phacoemulsification - foldable intra-ocular lens surgery with injector)

Exclusion Criteria:

1. Combined surgery
2. Previous intraocular surgery
3. Previous corneal refractive surgeries less than 6 months before screening
4. Non Senile or non pre-senilecataract (e.g.: traumatic, pathological or congenital cataract)
5. Pupillary abnormalities (irregular, etc.)
6. Iris synechiae
7. Eye movement disorder (nystagmus, etc.)
8. Dacryocystitis and all other pathologies of tears drainage system
9. History of Inflammatory ocular disease (Iritis, uveitis, herpetic keratitis)
10. Corneal, epithelial, stromal or endothelial, residual or evolutionary disease (including corneal ulceration and superficial punctuate keratitis)
11. History of ocular traumatism, infection or inflammation within the last 3 months
12. Pseudo-exfoliation, exfoliative syndrome
13. Prior intravitreal injections within 7 days of the surgery
14. IOP over 25mmHg under treatment
15. Best corrected visual acuity < 1/10
16. Patient already included in the study for phakoexeresis
17. History of ophthalmic surgical complication (cystoid macular oedema, etc.)
18. Diabetes mellitus
19. Surdity
20. Pakinsondisease
21. Excessive anxiety
22. Any other medical or surgical history, disorder or disease such as acute or chronic severe organic disease: hepatic, endocrine neoplasic, hematological diseases, severe psychiatric illness, relevant cardiovascular abnormalities (such as unstable angina, bradycardia, atrial fibrillation,uncontrolled hypertension: systolic blood pressure over 140 mm Hg, diastolic blood pressure over 90 mmHg) and/or any complicating factor or structural abnormality judged by the investigator to be incompatible with the study.
23. Known hypersensitivity to sulfonamides products or any of the components of the study medications or to test products Specific exclusion criteria for women
24. Pregnancy (positive pregnancy test), lactation
25. Women of childbearing potential without an acceptable effective method of contraception (oral contraceptive, intra-uterine device, subcutaneous contraceptive implant) until end of the study participation OR
26. Women not hysterectomized, not menopaused nor surgically sterilized. Exclusion criteria related to general conditions
27. Inability of patient and/or relatives to understand the study procedures and thus inability to give informed consent
28. Non-compliant patient and/or relatives (e.g. not willing to attend the follow-up visits, way of life interfering with compliance)
29. Participation in anotherclinicalstudy
30. Already included once in this study
31. Ward of court
32. Patient not covered by the Social Security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Alio, MD, Principal Investigator — Vissum Alicante, Calle del Cabañal 1, 03016 Alicante, Spain
Locations (27):
- Italy (16):
  - Policlinico S. Orsola-Malpighi - Dipartimento testa collo, U.O. Oftalmologia Ciardella, Bologna
  - A.O. Mater Domini di Catanzaro - U.O. Oculistica, Catanzaro
  - A.O.U. Careggi di Firenze - Dipartimento neuromuscoloscheletrico e organi di senso, reparto di oculistica, Florence
  - "IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano" - Dipartimento di chirurgia, U.O. Oculistica, Milan
  - Gruppo Multimedica Ospedale San Giuseppe di Milano - Clinica oculistica, Milan
  - Ospedale San Raffaele IRCCS - Clinica oculistica, Milan
  - ASST Santi Paolo e Carlo - Presidio Ospedale San Paolo - Dipartimento testa collo, reparto di oculistica, Milan
  - Fondazione IRCCS Policlinico S. Matteo - Dipartimento di scienze chirurgiche, U.O. Oculistica, Pavia
  - A.O. di Perugia - Ospedale S. Maria della Misericordia di Perugia - Clinica oculistica, Perugia
  - A.O.U. Pisana - Cisanello - D.A.I. Specialità chirurgiche, U.O. Oculistica, Pisa
  - Policlinico Universitario Campus Bio-medico di Roma - U.O.C. Oftalmologia, Roma
  - Fondazione PTV Policlinico Tor Vergata - Dipartimento benessere della salute mentale e neurologica, dentale e degli organi di senso, U.O.S.D. Oculistica, Roma
  - Ospedale Oftalmico di Roma (ASL Roma 1) - Dipartimento di oculistica e rete oftalmologica, Roma
  - IRCCS Fondazione G.B. Bietti di Roma - U.O.S. Segmento anteriore con annessi oculari, Roma
  - A.O.U. Senese - Università degli Studi di Siena - Dipartimento della salute mentale e degli organi di senso, U.O.C. Oculistica, Siena
  - Az. Sanitaria Universitaria Integrata di Udine - P.O. Universitario "Santa Maria della Misericordia" - Dipartimento di chirurgia specialistica, clinica oculistica, Udine
- Slovakia (8):
  - Izak Vision Center s.r.o., Banská Bystrica
  - FNsP F. D. Roosevelta Banská Bystrica II. Očná klinika SZU, Banská Bystrica
  - ROBIN LOOK spol. s r.o., Centrum mikrochirurgie oka, Bratislava
  - Vesely Očná Klinika, s.r.o., Bratislava
  - 3F s.r.o. Očná ambulancia a optika, Košice
  - UVEA KLINIKA, s.r.o., Martin
  - VIDISSIMO s. r. o. Očná klinika, Trenčín
  - Fakultná nemocnica s poliklinikou Žilina Očné oddelenie, Žilina
- Spain (3):
  - Oftalvist Cio Jerez Clinic, Jerez de la Frontera, Cadiz
  - Vissum alicante, Alicante
  - Instituto Oftalmológico Integral Servicio de Oftalmología Admiravisión en Clínica Corachan, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Figus M, Giansanti F, Villani E, Alio JL, Janco L, Mercuri S, Camnasio S, Cagini C. Chloroprocaine 3% Gel as a Novel Ocular Topical Anesthetic: Results from a Multicenter, Randomized Clinical Trial in Patients Undergoing Cataract Surgery. J Ocul Pharmacol Ther. 2024 Mar;40(2):117-125. doi: 10.1089/jop.2023.0096. PMID 38489057

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 410 subjects were screened in the study, 64 of which were dropped as screen failure and 346 were randomised to receive a treatment. From the 346 subjects randomised, 338 were treated and received the drug that was assigned at the randomization procedure, while 8 discontinued before treatment. Eventually, 335 subjects completed the study since discontinuation issues occurred for three subjects, one due to an AE and two lost to follow-up
Groups:
- Chloroprocaine 3%: All the eligible patients will be administrated by Chloroprocaine 3 % according to the randomization criteria.
  Chloroprocaine 3%: Administration: three IMP drops instillation as follow:
  * 1st Drop instillation, then wait for 5 minutes
  * Eye Disinfection, then wait for 2 minutes
  * 2nd Drop instillation, then wait for 1 minute
  * 3rdDrop instillation, then wait for 1 minute
  * Start of Surgery.
- Tetracaine 0.5%: All the eligible patients will be administrated by Tetracaine 0.5% according to the randomization criteria.
  Tetracaine 0.5%: Administration: three IMP drops instillation as follow:
  * 1st Drop instillation, then wait for 5 minutes
  * Eye Disinfection, then wait for 2 minutes
  * 2nd Drop instillation, then wait for 1 minute
  * 3rdDrop instillation, then wait for 1 minute
  * Start of Surgery.
Period: Overall Study
Arm/Group | Chloroprocaine 3% | Tetracaine 0.5%
Started | 167 | 171
Completed | 167 | 168
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chloroprocaine 3% | Tetracaine 0.5% | Total
Number analyzed (Participants) | 167 | 171 | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (10.3) | 68.8 (9.9) | 69.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 86 | 180
  Male | 73 | 85 | 158
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Each Treatment Group With a Successful Surface Anesthesia
Description: Τhe primary endpoint is the number of partecipants in each treatment group with a successful surface anesthesia, without any supplementation at the time point T4 (1 minute after the 3rd drop installation)
Time Frame: Before Intra Ocular Lens (IOL) implantation surgery.
Measure: Number; unit: participants
Arm/Group | Chloroprocaine 3% | Tetracaine 0.5%
Number analyzed (Participants) | 167 | 171
participants
  Anesthesia Success | 153 | 152
  Anesthesia NO Success | 14 | 19

2. Secondary Outcome: Changes in Ocular Symptoms
Description: Changes in ocular symptoms (pain, irritation/burning/stinging, foreign body sensation) will be graded by the patients according to the following scale (0 is the minimum value and 3 is tha maximum value) (0 = absent, 1 = mild, 2 = moderate, 3 = severe) during the study on Visit 1-selection and on visit 4-final
Time Frame: Visit 1 (Day -90/Day -1) and Visit 4 (Day 8 ± 1 day), up to approximately 102 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chloroprocaine 3% | Tetracaine 0.5%
Number analyzed (Participants) | 167 | 171
score on a scale
  Foreign Body Sensation visit1 | 0.08 (0.32) | 0.06 (0.33)
  Foreign Body Sensation visit4 | 0.19 (0.43) | 0.17 (0.41)
  Irritation/Burning/Stinging visit1 | 0.11 (0.33) | 0.11 (0.37)
  Irritation/Burning/Stinging visit4 | 0.11 (0.36) | 0.15 (0.39)
  pain visit1 | 0.01 (0.11) | 0.01 (0.08)
  pain visit4 | 0.05 (0.24) | 0.05 (0.24)

3. Secondary Outcome: Objective Ocular Signs
Description: - Objective ocular signs assessed by slit lamp examination, flare, and other objective ocular signs will be graded according to the following scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe. The minimum value is 0 and maximum value is 3
Time Frame: Visit 1 (Day -90/Day -1) and Visit 4 (Day 8 ± 1 day), up to approximately 102 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chloroprocaine 3% | Tetracaine 0.5%
Number analyzed (Participants) | 167 | 171
score on a scale
  Anterior Chamber Cells and Flare visit1 | 0 (0) | 0 (0)
  Anterior Chamber Cells and Flare visit4 | 0.04 (0.24) | 0.03 (0.2)
  Chemosis visit1 | 0.03 (0.17) | 0.04 (0.23)
  Chemosis visit4 | 0.09 (0.33) | 0.09 (0.33)

4. Secondary Outcome: Fluoresceine
Description: Modification of the basal status evaluated with fluorescein test Approximately 2-3 minutes following fluorescein instillation, corneal staining was to be evaluated in both eyes, using a slit lamp, based on the Oxford scale (grades of 0-5: 0 is normal, 5 is severe abnormal).
Time Frame: Visit 1 (Day -90/Day -1) and Visit 4 (Day 8 ± 1 day), up to approximately 102 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chloroprocaine 3% | Tetracaine 0.5%
Number analyzed (Participants) | 167 | 171
score on a scale
  Corneal Fluorescein Staining visit1 | 0.21 (0.61) | 0.16 (0.52)
  Corneal Fluorescein Staining visit4 | 0.32 (0.68) | 0.25 (0.66)

5. Secondary Outcome: Endothelial Cell Counts
Description: Modification of the basal status of the Endothelial cell counts evaluated with the specular microscopy
Time Frame: Visit 1 (Day -90/Day -1) and Visit 4 (Day 8 ± 1 day), up to approximately 102 days
Measure: Mean (Standard Deviation); unit: cell/mm^2
Arm/Group | Chloroprocaine 3% | Tetracaine 0.5%
Number analyzed (Participants) | 167 | 171
cell/mm^2
  Endothelial Cells Count [cell/mm2] visit1 | 2440.76 (378) | 2511.89 (325.32)
  Endothelial Cells Count [cell/mm2] visit4 | 2049.88 (620.43) | 2166.96 (517.41)

6. Secondary Outcome: Corneal Thickness
Description: Modification of the basal status of the assesment (Corneal thickness). Measurement of the central corneal thickness was to be performed with a pachymeter
Time Frame: Visit 1 (Day -90/Day -1) and Visit 4 (Day 8 ± 1 day), up to approximately 102 days
Measure: Mean (Standard Deviation); unit: um
Arm/Group | Chloroprocaine 3% | Tetracaine 0.5%
Number analyzed (Participants) | 167 | 171
um
  visit 1 (Day -90/Day -1) | 539.59 (39.3) | 536.59 (37.16)
  visit 4 (Day 8 ± 1 day) | 557.8 (48.8) | 546.54 (42.15)

7. Secondary Outcome: Best Far Corrected Visual Acuity
Description: Modification of the basal status of the assesment evaluated by LogMAR (Logarithm of the Minimum Angle of Resolution). When using a LogMAR chart, visual acuity is scored with reference to the logarithm of the minimum angle of resolution, as the chart's name suggests. An observer who can resolve details as small as 1 minute of visual angle scores LogMAR 0, since the base-10 logarithm of 1 is 0; an observer who can resolve details as small as 2 minutes of visual angle (i.e., reduced acuity) scores LogMAR 0.3, since the base-10 logarithm of 2 is near-approximately 0.3; and so on.
Time Frame: Visit 1 (Day -90/Day -1) and Visit 4 (Day 8 ± 1 day), up to approximately 102 days
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Chloroprocaine 3% | Tetracaine 0.5%
Number analyzed (Participants) | 167 | 171
LogMAR
  Best Corrected Visual Acuity LogMAR visit1 | 0.49 (0.31) | 0.47 (0.32)
  Best Corrected Visual Acuity LogMAR visit4 | 0.12 (0.19) | 0.08 (0.15)

8. Secondary Outcome: Number of Participants With Abnormalities of the Retina, Macula, or Optic Nerve by Fundoscopy
Description: Modification of the basal status of the assesment. Dilated fundus examination on retina, macula, optic nerve.
Time Frame: Visit 1 (Day -90/Day -1) and Visit 4 (Day 8 ± 1 day), up to approximately 102 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroprocaine 3% | Tetracaine 0.5%
Number analyzed (Participants) | 167 | 171
Participants
  macula abnormal V1 | 15 | 16
  macula abnormal V4 | 13 | 10
  optic nerve abnormal V1 | 16 | 16
  optic nerve abnormal V4 | 12 | 10
  retina abnormal V1 | 13 | 11
  retina abnormal V4 | 13 | 12

9. Secondary Outcome: Intra-ocular Pressure
Description: Modification of the basal status of the assesment. Intraocular pressure (in mmHg) was assessed according to site current practice (air puff or applanation tonometer).
Time Frame: Visit 1 (Day -90/Day -1) and Visit 4 (Day 8 ± 1 day), up to approximately 102 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Chloroprocaine 3% | Tetracaine 0.5%
Number analyzed (Participants) | 167 | 171
mmHg
  visit 1 Selection | 15 (2.69) | 15 (2.46)
  visit 4 Final | 14.7 (2.8) | 14.88 (3.05)

10. Secondary Outcome: Surgeon Satisfaction
Description: Evaluation of surgeon satisfaction. Surgeon satisfaction was assessed through the question "How do you consider the study product global tolerance?", at a scale (a score of 0 is the minimum value with the best outcome and 3 is the maximum value with the worst outcome): (0) Very satisfactory, (1) Satisfactory, (2) Not very satisfactory, (3) Unsatisfactory. It is recorded at V2 and filled in by the surgeon who had performed the study. It is measured at Visit 2.
Time Frame: day 1 - visit2 (Inclusion visit/Surgery)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chloroprocaine 3% | Tetracaine 0.5%
Number analyzed (Participants) | 167 | 171
score on a scale | 0.17 (0.41) | 0.17 (0.47)

11. Secondary Outcome: Patient Global Satisfaction
Description: Patient global satisfaction at D1 based on a 5-question questionnaire read by a masked observer.
  A question read by a masked observer assessed the patient satisfaction about the overall anesthesia during the surgery: "Overall, how satisfied are you with the topical study product used for your local anesthesia during your cataract surgery?" It was measured with 5 possible answers (Likert satisfaction scale): Very satisfied (0), Globally satisfied (1), Neither satisfied nor Unsatisfied (2), Globally unsatisfied (3), Very unsatisfied (4). It was measured at Visit 3.
Time Frame: day 1 - visit2 (Inclusion visit/Surgery) after the treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chloroprocaine 3% | Tetracaine 0.5%
Number analyzed (Participants) | 167 | 171
score on a scale | 1.35 (0.66) | 1.27 (0.52)

ADVERSE EVENTS:
Time Frame: Adverse events were to be monitored throughout the course of the study Visit 1 (Day -90/Day -1) and Visit 4 (Day 8 ± 1 day)) up to "Visit 5 (Day 28 ± 3 days; approximately 129 days
Description: Any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with treatment
Arm/Group | Chloroprocaine 3% | Tetracaine 0.5%
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/171
Serious Adverse Events (participants affected / at risk) | 0/167 | 0/171
Other Adverse Events (participants affected / at risk) | 14/167 | 19/171
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chloroprocaine 3% (N=167) | Tetracaine 0.5% (N=171)
corneal Dystrophy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Conjunctival hemorrhage (Eye disorders) | 1 (1) | 0 (0)
congiunctivitis (Eye disorders) | 0 (0) | 1 (1)
corneal degeneration (Eye disorders) | 0 (0) | 1 (1)
cornela disorder (Eye disorders) | 0 (0) | 1 (1)
corneal edema (Eye disorders) | 5 (5) | 2 (2)
eye discharge (Eye disorders) | 0 (0) | 1 (1)
hyperesthesia (Eye disorders) | 1 (1) | 0 (0)
iridocele (Eye disorders) | 0 (0) | 1 (1)
lens dislocation (Eye disorders) | 0 (0) | 1 (1)
ocular Hypertension (Eye disorders) | 0 (0) | 1 (1)
photophobia (Eye disorders) | 1 (1) | 1 (1)
keratitis (Eye disorders) | 1 (1) | 1 (1)
deformity (Eye disorders) | 0 (0) | 1 (1)
pupillary disorder (Eye disorders) | 0 (0) | 1 (1)
Retinal pigment epitheliopathy (Eye disorders) | 1 (1) | 0 (0)
general disorder (Eye disorders) | 2 (2) | 0 (0)
pyrexia (Eye disorders) | 1 (1) | 0 (0)
Sensation of foreign body (Eye disorders) | 1 (1) | 0 (0)
edema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
blood pressure increased (Investigations) | 0 (0) | 3 (3)
Intraocular pressure increased (Investigations) | 1 (1) | 3 (6)
trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
devise dislocation (Product Issues) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT04685538/Prot_SAP_000.pdf